CLINICAL TRIAL: NCT04087148
Title: Linear Growth of Children With Congenital Adrenal Hyperplasia.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali Hussin Mohamed, principal Investigator, Assiut University
Other Study IDs: GCAH
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Congenital Adrenal Hyperplasia
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients: patients who were diagnosed as having CAH of at least 1 y duration. and On glucocorticoid replacement therapy .
- controls: A comparable number of age and sex matched apparently normal children will be included as control.

SUMMARY:
The congenital adrenal hyperplasias (CAHs) comprise a family of autosomal recessive disorders that disrupt adrenal steroidogenesis. Three specific enzyme deficiencies are associated with virilization of affected women. The most common form is 21-hydroxylase deficiency (21-OHD) due to mutations in the 21-hydroxylase (CYP21A2) gene. Other virilizing forms include 3b-hydroxysteroid dehydrogenase type 2 (HSD3B2) and 11b-hydroxylase deficiencies associated with mutations in the HSD3B2 and 11b-hydroxylase (CYP11B1) genes, respectively.

DETAILED DESCRIPTION:
It has been reported that approximately one child in every 18000 born in Great Britain has CAH. In North America, the incidence varies from 1:15000 to 1:16000. The reported rates of CAH have been as high as 1:280 among the Yupik people of Alaska and 1:2100 on the French island of Réunion in Indian ocean; both of these populations are geographically isolated. The reported incidence of CAH in the two Brazilian states that have routinely included CAH in their public newborn screening programs is 1:11655 in the South (Santa Catarina) and 1:10325 in Midwest (Goiás).

Salt-losing CAH accounts for about three quartes of cases reported and non-salt losing CAH for one quarter. Non-classic is more common ;Estimated as 1 in 1000-2000 in white populations. It is more frequent in certain ethnic groups, such as the Ashkenazi Jewish population. The mild non-classic form is a common cause of hyperandrogenism.

Treatment of classic 21-OHD consists of replacement doses of gluco- (GC) and mineralocorticoids aiming to reduce excess androgen, and to allow adequate linear growth. However, several series report that growth in these children is below expectation, as compared with both the reference population and the target height (TH).

The reasons for the inadequate growth and impairment of the final height (FH) are not completely understood. A major cause is the difficulty in accomplishing a fine balance between inhibition of excess androgen production which accelerates bone maturation and adequate GC replacement itself which even at slightly supraphysiologic doses can be deleterious to growth.

ELIGIBILITY:
Inclusion criteria:

* Age: 1-18 y.
* Both sexes.
* All patients who were diagnosed as having CAH of at least 1 y duration.
* On glucocorticoid replacement therapy .

Exclusion criteria:

* Patients diagnosed as CAH for less than 1 year duration.
* Patients with deficient data at the time of diagnosis.
* Patients missed for follow up.
* Syndromatic patients.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: • pediatric patients with congenital adrenal hyperplasia who are taking glucocorticoid replacement therapy and attending Endocrine unit of Assiut University Children Hospital within one year.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-09-24 (Estimated); Primary Completion 2020-10-24 (Estimated); Study Completion 2021-10-24 (Estimated)

PRIMARY OUTCOMES:
factors affecting linear growth in children with CAH. | 6 months
  by using appropriate growth charts and doing follow up wrist x-ray .

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Delle Piane L, Rinaudo PF, Miller WL. 150 years of congenital adrenal hyperplasia: translation and commentary of De Crecchio's classic paper from 1865. Endocrinology. 2015 Apr;156(4):1210-7. doi: 10.1210/en.2014-1879. Epub 2015 Jan 30. PMID 25635623
- [Background] Silveira EL, dos Santos EP, Bachega TA, van der Linden Nader I, Gross JL, Elnecave RH. The actual incidence of congenital adrenal hyperplasia in Brazil may not be as high as inferred--an estimate based on a public neonatal screening program in the state of Goias. J Pediatr Endocrinol Metab. 2008 May;21(5):455-60. doi: 10.1515/jpem.2008.21.5.455. PMID 18655527
- [Background] Nunes AK, Wachholz RG, Rover MR, Souza LC. [Prevalence of disorders detected by newborn screening in Santa Catarina]. Arq Bras Endocrinol Metabol. 2013 Jul;57(5):360-7. doi: 10.1590/s0004-27302013000500005. Portuguese. PMID 23896802
- [Background] Trapp CM, Oberfield SE. Recommendations for treatment of nonclassic congenital adrenal hyperplasia (NCCAH): an update. Steroids. 2012 Mar 10;77(4):342-6. doi: 10.1016/j.steroids.2011.12.009. Epub 2011 Dec 13. PMID 22186144
- [Background] Nebesio TD, Eugster EA. Growth and reproductive outcomes in congenital adrenal hyperplasia. Int J Pediatr Endocrinol. 2010;2010:298937. doi: 10.1155/2010/298937. Epub 2010 Feb 1. PMID 20148087